CLINICAL TRIAL: NCT06514586
Title: The Efficacy of Topical Vaginal Oxytocin Gel in Postmenopausal Women With Vuluvovaginal Atrophy: A Randomized Controlled Trial
Brief Title: The Efficacy of Topical Vaginal Oxytocin Gel in Postmenopausal Women With Vulvovaginal Atrophy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oxagon (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Oxagon
Record Dates: First submitted 2024-04-22; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Vaginal Atrophy; Genitourinary Syndrome of Menopause; Vulvar Atrophy
Keywords: vulvovaginal atrophy; postmenopause; vulvovaginal; atrophy
MeSH Terms: conditions — Atrophy | interventions — Oxytocin; Hypromellose Derivatives

STUDY DESIGN:
Intervention Model Description: A Double-Blinded Randomized Controlled Trial The study includes 2 arms. The subjects will be randomized to receive (apply) either oxytocin topical gel (intervention arm) or placebo gel (control arm).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MenOxy (Active Comparator): The investigational product will contain a Plastic tube containing 36 g of study product (gel) and a Vaginal calibrated plastic applicator for dose (1 ml) administration. The active constituent is oxytocin 600 IU/ml dissolved in a gel based on Hypromellose with a pH of 3.8.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): The placebo gel will match the IP gel (Hypromellose) with a pH of 3.8, without oxytocin.
  Interventions: Other: Hydroxypropyl methylcellulose

INTERVENTIONS:
Drug: Oxytocin — Oxytocin gel 600 IU . 1mg/g
  Arms: MenOxy
Other: Hydroxypropyl methylcellulose — Placebo
  Arms: Placebo

SUMMARY:
A Phase three randomized, double-blinded, study to asses the efficacy and safety of oxytocin gel in postmenopausal women with vaginal atrophy due to Genitourinary Syndrome of Menopause GSM.

DETAILED DESCRIPTION:
A Phase three randomized, double-blinded, placebo- controlled study to asses the efficacy and safety of oxytocin gel in postmenopausal women with vaginal atrophy due to Genitourinary Syndrome of Menopause GSM. This study shall include 242 subjects. After screening , subject who meet eligibility criterial will be randomized in a 1:1 ratio to receive wither study intervention or placebo to be applied once daily for sixty days and followed up extra fifteen days. objectives is to evaluate the efficacy and effectiveness of topical oxytocin gel compared with placebo in improving postmenopausal vaginal atrophy symptoms in women with GSM , also assessing the safety and tolerability of topical oxytocin gel.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal, sexually active female subject of age 47 - 65 years, at the time of randomization, willing to provide an informed consent.
2. Physical Assessment showing vaginal atrophy (according to the following criteria: pale, smooth, or shiny vaginal epithelium, friable, epithelium showing no rugae, loss of elasticity or turgor of the skin, dryness of labia, fusion of labia minora, vulvar lesions, or erythema.) 3. Patients with at least one present symptom (ex. vaginal dryness, itching, burning, dysuria, and/or dyspareunia) and able to identify one symptom as the most bothersome symptom, with at least moderate severity.

4. Vaginal smear cytology at screening showing ≤ 5% superficial cells 5. Vaginal pH > 5.0 at screening 6. A level of estradiol ≤ 30 pg/mL and a level of Follicle Stimulating Hormone (FSH) > 40 milli International Units (mIU)/ml at screening 7. Be willing to abstain from sexual activity and the use of vaginal douching within 24 hours prior to vaginal pH measurements at screening and the study follow-up visits

Exclusion Criteria:

1. Previous treatment with other local non-hormonal moisturizers/hormonal products within 1 month or use of lubricants within 1 week prior to inclusion.
2. Women taking systemic hormone replacement or pills within the last 6 months.
3. Current or history of endometrial hyperplasia or uterine/endometrial, breast, or ovarian cancer, or undiagnosed vaginal bleeding
4. Any untreated urogenital infection within 14 days prior to randomization.
5. Ongoing treatment with systemic medications for other non-related health conditions which might impact the study results and have the potential to bring about change in the vaginal environment e.g. glucocorticosteroids, antibiotics, etc.
6. Critically ill patients.
7. Patients with severe renal impairment (GFR < 30 ml/min/1.73 m2 as measured by the Cockcroft-Gault formula).
8. Patients with known severe hepatic impairment (Child-Pugh C; 10 - 15 points), biliary cirrhosis, or cholestasis.
9. Patients with known or suspected allergy or any contraindications to oxytocin.

Ages: 47 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The mean change from the baseline to Day 60 of the severity of the Most Bothersome Symptom (MBS) self-assessment. | 60 days
  MBS is a moderate to severe symptom identified as the most bothersome by the subject at baseline, recorded as none, mild, moderate, or severe was analyzed using the score values of 0, 1, 2, or 3, respectively. Symptoms include vaginal dryness, vaginal/vulvar irritation/itching, dysuria, vaginal pain (dyspareunia), or bleeding associated with sexual activity.
The mean change from the baseline to Day 60 of the vaginal pH | 60 days
  Vaginal pH as measured by a pH strip applied directly to the lateral wall of the vagina, recording the pH value (to one decimal) according to the comparison to the color chart.
The mean change from the baseline to Day 60 of the Vaginal Maturation Index (VMI) | 60 days
  VMI is calculated using the Meisels'(Meisels, 1967) formula: (0 * Parabasal Cells) + (0.5 * Intermediate Cells) + (1 * Superficial Cells).

SECONDARY OUTCOMES:
The mean changes in MBS severity, pH, and VMI from the baseline to Days 30 and 75 | Days 30 and 75
The percentage of subjects identified as Responders on days 60 and 75. | Days 60 and 75
  A responder is a subject meeting all the following criteria: at least 1 point improvement (decrease) in the severity of the MBS, at least a 0.5-point decrease in the vaginal pH, and at least 20% improvement in the VMI.
The mean change from the baseline to Days 30, 60, and 75 of the physical examination of the vulva and vagina | Days 30, 60, and 75
  Assessment of the physical signs of VA (Vaginal secretions, Vaginal Epithelial Integrity, Vaginal Epithelial Surface Thickness, and Vaginal Color) as evaluated by the physician/gynecologist and corresponding to none, mild, moderate, or severe atrophy and analyzed using the score values of 0, 1, 2, and 3, respectively.
The mean changes from the baseline to Days 30, 60, and 75 in Vaginal Wall Thickness as measured by transvaginal ultrasound. | Days 30, 60, and 75
The mean changes from the baseline to Days 30, 60, and 75 in Doppler indices measured by transvaginal ultrasound. | Days 30, 60, and 75
The mean change from the baseline to Days 60 and 75 in selected items from the Female Sexual Function Index (FSFI). | Days 60, and 75
The mean change from the baseline to Days 60 and 75 in patient-reported psychometric outcomes. | Days 60 and 75
The number and percentage of subjects on Days 30, 60, and 75 reporting Treatment-Emergent Adverse Event (TEAE), defined as any AE that occurs on or after the application of the first dose of the study intervention. | Days 30, 60 and 75
The rate of abnormal findings on Days 30, 60, and 75 during the physical, gynecological, and breast examinations. | Days 30, 60 and 75
The rate of abnormal findings on Days 30, 60, and 75 of the transvaginal ultrasound for women with an intact uterus only. | Days 30, 60 and 75
The mean medication incompliance rate (%) will be calculated in Days 30, and 60 for each subject as [(Total number of missed doses) / (Expected number of applications)] *100%. | Days 30,and 60
The incidence of AEs reported by the subjects, summarized by system organ class, severity, and relationship to study intervention, over the course of treatment. | Days 30, 60 and 75

OTHER OUTCOMES:
The mean change in weight from baseline to days 60 and 75, and BMI from baseline to day 75. | Days 60 and 75
The number of subjects reporting changes in appetite (satiety/hunger) on days 30, 60, and 75. | Days 30, 60 and 75
The mean change in fasting blood glucose, HbA1C, and insulin levels from baseline to days 60. | Day 60
The mean change in blood pressure from baseline to days 30, 60, and 75. | Days 30, 60 and 75
The mean change in IL-6 from baseline to days 60. | Day 60
The mean changes in metabolic bone marker (Alkaline phosphatase (ALP)) from baseline to day 60 | Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Assem Anwar, Principal Investigator — Azhar Univeristy
Locations (1):
- Oxagon, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided